CLINICAL TRIAL: NCT07371052
Title: Effects of Short-Term Olive Leaf Extract Supplementation in Elite Male Handball Players
Brief Title: Olive Leaf Extract in Handball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Büşra Demirer, Dr. Research Assistant, Nutritients, Karabuk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: handball players
Record Dates: First submitted 2026-01-15; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Handball Players
MeSH Terms: interventions — olive leaf extract

STUDY DESIGN:
Intervention Model Description: Parallel assigned
Who Masked: Participant, Care Provider, Investigator
Masking Description: double blind (participant investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): olive leaf extract supplemented
  Interventions: Dietary Supplement: Olive leaf extract
- Control group (Placebo Comparator): placebo capsule supplemented
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Olive leaf extract — OLE supplement (500 mg, standardized to 25% oleuropein)
  Arms: Study group
Other: Placebo — Sucrose capsules with the same color, scent, and size as OLE capsules.
  Arms: Control group

SUMMARY:
Olive leaf extract (OLE) is a natural supplement rich in phenolic compounds, especially oleuropein, which has antioxidant properties that may support recovery after physical exercise. While OLE has been studied for various health-related effects, its potential impact on exercise recovery and performance in elite athletes remains unclear.

This randomized, double-blind, placebo-controlled study was designed to evaluate the effects of four weeks of OLE supplementation on physical performance, sleep quality, and post-exercise muscle soreness in elite male handball players aged 18 to 25 years. Participants were randomly assigned to receive either a daily OLE supplement (500 mg, standardized to 25% oleuropein) or a placebo for four weeks. Physical performance, sleep quality, and muscle soreness were assessed at baseline, during the intervention, and at the end of the study period. Muscle soreness was additionally evaluated at 12 and 24 hours following exercise sessions.

ELIGIBILITY:
Inclusion Criteria:

* Male elite handball players aged 18 years or older
* Free from any diagnosed chronic disease, as determined by medical history
* Not following a calorie-restricted diet within the previous six months
* No use of nutritional supplements within the previous six months

Exclusion Criteria:

* Age under 18 years
* Smoking or alcohol consumption
* Presence of any diagnosed chronic disease
* Adherence to a regular calorie-restricted diet within the previous six months
* Use of nutritional supplements during the previous six months

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Muscle Soreness | Baseline, After intervention (two week later), After intervention (fourt week later)
  The severity of muscle soreness will be assessed using the Visual Analog Scale (VAS). Patients choose the appropriate score between 0 and 10. Higher scores indicate higher muscle soreness levels.
Squat jump height | Performance outcomes were assessed at baseline, week 2, and week 4 of the intervention period.
  Lower-body explosive performance was assessed using the squat jump test. Jump height was measured in centimeters (cm) with higher values indicating better explosive performance.
Peak anaerobic power | baseline, week 2, and week 4.
  Peak anaerobic power was assessed using the Wingate anaerobic test. Peak power output was recorded in watts (W) during the 30-second maximal cycling test. Higher values indicate greater anaerobic power.
Countermovement jump height | Assessments were conducted at baseline, week 2, and week 4. Higher values indicate better explosive performance.
  Lower-body explosive performance was assessed using the countermovement jump test. Jump height was measured in centimeters (cm) with higher values indicating better explosive performance.
Mean anaerobic power | Baseline, week 2, and week 4
  Mean anaerobic power was assessed using the Wingate anaerobic test. Mean power output was calculated as the average power produced over the 30-second test and recorded in watts (W). Higher values indicate better anaerobic capacity.
Fatigue index | Baseline, week 2, and week 4
  Fatigue index was assessed using the Wingate anaerobic test and calculated as the percentage decline in power output from peak to minimum power during the 30-second test. Higher values indicate greater fatigue.

SECONDARY OUTCOMES:
Sleep quality | Total PSQI scores were recorded at baseline, week 2, and week 4 to evaluate changes in perceived sleep quality during the supplementation period.
  Sleep quality was assessed using the Pittsburgh Sleep Quality Index (PSQI) total score. The PSQI is a validated self-reported questionnaire consisting of 19 items, yielding a global score ranging from 0 to 21, with higher scores indicating poorer sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Karabuk University, Karabük, Central, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No